CLINICAL TRIAL: NCT04880759
Title: Pilot Study of Active Desk in Primary School : Effects on the Attention, Cognitive Capacities, Physical Capacities, Concentration and Well-being of Student and on the Classroom Climate
Brief Title: Pilot Study of Active Desk in Primary School : Effects on Cognitive Capacities, Physical Capacities and Well-being
Acronym: BICLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2021 DUCLOS; 2021-A00114-37 (Other: 2021-A00114-37)
Record Dates: First submitted 2021-04-14; First posted 2021-05-11 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cognition
Keywords: Cycling desk; Active workstation; Sedentary Behavior; Cognition; Child health; Body composition; Physical fitness
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bike desks in classroom (Experimental): All participants receive the same intervention: the use of bike desks during school.
  Interventions: Other: bike desks in the classroom

INTERVENTIONS:
Other: bike desks in the classroom — Children will use bike desks for 13 weeks during school time

SUMMARY:
Physical activity (PA) is insufficient in children with three quarters of them who do not meet the WHO's recommendations. Physical inactivity is growing during adolescence; in part due to the time spend in sedentary behaviors at school. The recent literature is highlighting the importance of physical activity on academic achievement, physical fitness and academic achievement in children. In addition, deleterious effects of sedentary behaviors have been demonstrated. At school, many strategies have been settled to break the prolonged sitting time. The use of workstations is one of them and allows to reduce sedentary time at school and increases physical activity without interrupting class. Active workstations like bike desks have demonstrated their effectiveness on physical activity but their effects have not been evaluated in primary school in France. In addition, few studies have evaluated the effects of bike desk use on the child's cognitive abilities.

The main objective of this project is to measure the variations linked to the use of bike desks (desk with pedals) for an average of 1h45mn per week (30min 3 to 4 times per week) for 13 weeks during school time in primary school pupils (aged 8 to 11 years) on the cognitive abilities (mental flexibility, working memory and inhibition) of children.

Our hypothesis is that the use of the bike desk for 1h45 per week will induce an increase in the attention and cognitive capacities (mental flexibility, working memory and inhibition) of the children. Other improvements that should be identified are the child's body composition, the classroom climate and the well-being of pupils and teachers. The children's physical capacities could also be increased, beyond what is expected given the normal evolution during the year.

DETAILED DESCRIPTION:
Two prospective schools have given their prior agreement : Sevigne Lafaye (Vichy) and Pierre Brossolette (Riom). The use of the bike desks in the classroom is part of the school project and will start at the same time as the study. There are 4 bike-desks in each class: 3 for the children and 1 for the teacher. Students pedaling during an overall of 13 weeks (7 weeks and 6 weeks) separated of one evaluation session week (T1). During weeks with evaluation sessions, children will not use bike desk. All children will therefore use the bike desks but only those who have signed the consent form.

An information meeting will be proposed in each school (visit 1). Then, subjects will have a pre-inclusion visit during a medical consultation where the eligibility criteria to participate in this study will be checked (visit 2). The children who have given their consent will have to participate in different evaluation sessions: baseline (T0), between to two pedaling sessions (T1) and at the end of the second session (T2). They are two parts of assessments for each session (T0, T1, T2):

* Cognitive test and the physical activity attraction test (visits 3, 5, 7)
* Body composition and physical capacity assessment (visits 4, 6, 8) Questionnaires will also be part of the assessment (T1 and T2).

ELIGIBILITY:
Inclusion Criteria:

* Children between 8 and 11 years old (inclusive)
* Girls and boys
* Children enrolled in CM1a and CM1b classes at the Pierre Brossolette school in Riom and in CM1/CM2 and CM2 classes at the Sévigné-Lafaye school in Vichy.
* Able to provide informed consent to research participation
* Registered in the French social security system

Exclusion Criteria:

* Medical or surgical history judged by the investigator to be incompatible with the study
* Any unstabilised chronic pathology
* Inability to pedal
* Inability or contraindication to physical activity
* Subjects with cardiorespiratory and/or osteoarticular disorders that limit their ability to perform physical tests or use the cycle desks
* Subjects with a progressive cardiovascular or neoplastic disease.
* Subjects with a major infection in the 3 months prior to inclusion
* Subject with chronic or acute inflammatory disease in the 3 months prior to inclusion
* Subject diagnosed and/or treated for schizophrenia, bipolar disorder, major depression
* Person under guardianship, curatorship or not subject to a social security scheme
* Refusal to sign written consent to participate by the participant or a parent or guardian

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Students cognitive abilities | Week 0
  Time to complete the Trail Making Test part A and B (seconds)
Students cognitive abilities | 7 weeks
  Time to complete the Trail Making Test part A and B (seconds)
Students cognitive abilities | 13 weeks
  Time to complete the Trail Making Test part A and B (seconds)

SECONDARY OUTCOMES:
Weight | Week 0
  Weight (kg) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan)
Body composition (body mass index) | Week 0
  Body mass index (kg/m^2) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan) by combining weight and height
Body composition (body fat mass) | Week 0
  Body fat mass (%) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan)
Weight | 7 weeks
  Weight (kg) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan)
Body composition (body mass index) | 7 weeks
  Body mass index (kg/m^2) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan) by combining weight and height
Body composition (body fat mass) | 7 weeks
  Body fat mass (%) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan)
Weight | 13 weeks
  Weight (kg) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan)
Body composition (body mass index) | 13 weeks
  Body mass index (kg/m^2) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan) by combining weight and height
Body composition (body fat mass) | 13 weeks
  Body fat mass (%) will be assessed by bioimpedance analysis with Tanita MC-780 (Tanita Corp., Tokyo, Japan)
Physical fitness (cardio-respiratory capacity) | Week 0
  Cardio-respiratory capacity will be assessed with 20 m shuttle test (ml.mn.kg-1)
Physical fitness (cardio-respiratory capacity) | 7 weeks
  Cardio-respiratory capacity will be assessed with 20 m shuttle test (ml.mn.kg-1)
Physical fitness (cardio-respiratory capacity) | 13 weeks
  Cardio-respiratory capacity will be assessed with 20 m shuttle test (ml.mn.kg-1)
Physical fitness (muscular strength) | Week 0
  Muscular strength will be assessed with Standing Broad Jump test (cm), Countermovement Jump test (cm) and Throw Medicine Ball test (cm)
Physical fitness (upper limbs muscular strength) | Week 0
  Muscular strength will be assessed with Handgrip test (kg)
Physical fitness (muscular strength) | 7 weeks
  Muscular strength will be assessed with Standing Broad Jump test (cm), Countermovement Jump test (cm) and Throw Medicine Ball test (cm)
Physical fitness (upper limbs muscular strength) | 7 weeks
  Muscular strength will be assessed with Handgrip test (kg)
Physical fitness (muscular strength) | 13 weeks
  Muscular strength will be assessed with Standing Broad Jump test (cm), Countermovement Jump test (cm) and Throw Medicine Ball test (cm)
Physical fitness (upper limbs muscular strength) | 13 weeks
  Muscular strength will be assessed with Handgrip test (kg)
Physical fitness (motor skills) | Week 0
  Motor skills will be assessed with the time to complete an obstacle course (seconds)
Physical fitness (motor skills) | 7 weeks
  Motor skills will be assessed with the time to complete an obstacle course (seconds)
Physical fitness (motor skills) | 13 weeks
  Motor skills will be assessed with the time to complete an obstacle course (seconds)
Implicit and explicit attraction to physical activity | Week 0
  Implicit and explicit attraction to physical activity will be assessed with Activity Preference Assessment (APA) computer test
Implicit and explicit attraction to physical activity | 7 weeks
  Implicit and explicit attraction to physical activity will be assessed with Activity Preference Assessment (APA) computer test
Implicit and explicit attraction to physical activity | 13 weeks
  Implicit and explicit attraction to physical activity will be assessed with Activity Preference Assessment (APA) computer test
Teachers' perceptions of students' well-being | Week 0
  Questionnaire created by the National Education. Items will be rated from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Teachers' perceptions of students' well-being | 7 weeks
  Questionnaire created by the National Education. Items will be rated from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Teachers' perceptions of students' well-being | 13 weeks
  Questionnaire created by the National Education. Items will be rated from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Students and teachers' perceived well-being | 7 weeks
  Questionnaire created by the National Education. Items will be rated with smiley or rating from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Students and teachers' perceived well-being | 13 weeks
  Questionnaire created by the National Education. Items will be rated with smiley or rating from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Classroom climate/atmosphere | 7 weeks
  Questionnaire created by the National Education. Items will be rated from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Classroom climate/atmosphere | 13 weeks
  Questionnaire created by the National Education. Items will be rated from 1 to 5: 1 unsatisfactory; 2 marginally satisfactory; 3 neutral; 4 satisfactory; 5 very satisfactory. Higher scores mean a better outcome.
Possible factors of failure of the strategy | 13 weeks
  Questionnaire: socioeconomical level of parents, reason for refusal to participate , parents feeling, students feeling, teachers feeling. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France